CLINICAL TRIAL: NCT01696539
Title: Pilot Intervention Study of the Impact of Sustainable Daily Physical Activity on Health and Quality of Life in a Cohort of Men With Prostate Cancer in Sweden: Steps for PRosTAte Cancer Health and Survival (SPaRTACuS)
Brief Title: Steps for PRosTAte Cancer Health and Survival (SPaRTACuS): Pilot Study of a Walking Intervention to Improve Health and Quality of Life in Prostate Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Ove Andrén, Associate Professor and Chair of Urology, Örebro University, Sweden
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Spartacus01
Record Dates: First submitted 2012-09-16; First posted 2012-10-01 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Prostatic Neoplasm
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Walking Intervention (Experimental): Participants are provided with the current standard of prostate cancer care, and are additionally encouraged to walk 10,000 steps per day, as measured by pedometers provided at start of intervention. Once a week, participants will take part in a group walk with 7-8 other participants and a research nurse. Participants are also encouraged to keep a walking journal, in which they record the number of steps they walk each day. This journal is submitted to investigators at the end of the intervention period.
  Interventions: Behavioral: Walking Intervention
- Standard of Care (Active Comparator): Participants are provided with the current standard of prostate cancer care, but are not assigned to a physical activity intervention.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: Walking Intervention — Participants are provided with the current standard of prostate cancer care, and are additionally encouraged to walk 10,000 steps per day, as measured by pedometers provided at start of intervention. Once a week, participants will take part in a group walk with 7-8 other participants and a research nurse. Participants are also encouraged to keep a walking journal, in which they record the number of steps they walk each day. This journal is submitted to investigators at the end of the intervention period.
  Arms: Walking Intervention
Other: Standard of Care — Participants are provided with the current standard of prostate cancer care, but are not assigned to a physical activity intervention.
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to determine whether sustainable daily physical activity is effective in improving biological indicators of health and self-reported quality of life in men with prostate cancer.

DETAILED DESCRIPTION:
Living with prostate cancer is a unique challenge faced by millions of men across the globe. Existing research has indicated many potential methods of attenuating prostate cancer progression and preserving patients' quality of life, but is lacking in definitive conclusions regarding the effectiveness of these methods in practice. This study seeks to further investigate the impact of post-diagnosis physical activity on biological indicators of health and self-reported quality of life in a cohort of men with prostate cancer in Sweden. Participants are randomized to either a walking intervention group, which encourages walking 10,000 steps per day for one year, or to a standard-or-care control group, and followed for 11 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 80 years or younger
* Histologic confirmation of prostate cancer
* Clinically or pathologically staged as locally advanced or early metastatic prostate cancer
* Diagnosis within 1 year of study enrollment
* Willing and able to walk 10,000 steps per day

Exclusion Criteria:

* Age greater than 80 years old at enrollment
* Inability to understand the language spoken in host country
* Physically unable to walk 100 meters unassisted
* Diagnosed with dementia or severe psychiatric disease
* Any prior cancer diagnosis
* Has experienced a myocardial infarction or stroke within six months of cancer diagnosis

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

SECONDARY OUTCOMES:
C-Reactive Protein | At time of randomisation(March 1, 2010) and after 11 weeks
  Levels assessed in blood. Blood draw performed by clinician at start and 11 weeks after start of intervention.
High-Density Lipoprotein | At time of randomisation(March 1, 2010) and after 11 weeks
  Levels assessed in blood. Blood draw performed by clinician at start and 11 weeks after start of intervention.
Adiponectin | At time of randomisation(March 1, 2010) and after 11 weeks
  Levels assessed in blood. Blood draw performed by clinician at start and 11 weeks after start of intervention.
Total Cholesterol | At time of randomisation(March 1, 2010) and after 11 weeks
  Levels assessed in blood. Blood draw performed by clinician at start and 11 weeks after start of intervention.
Triglycerides | At time of randomisation(March 1, 2010) and after 11 weeks
  Levels assessed in blood. Blood draw performed by clinician at start and 11 weeks after start of intervention.
Insulin | At time of randomisation(March 1, 2010) and after 11 weeks
  Levels assessed in blood. Blood draw performed by clinician at start and 11 weeks after start of intervention.
Testosterone | At time of randomisation(March 1, 2010) and after 11 weeks
  Levels assessed in blood. Blood draw performed by clinician at start and 11 weeks after start of intervention.
Estradiol | At time of randomisation(March 1, 2010) and after 11 weeks
  Levels assessed in blood. Blood draw performed by clinician at start and 11 weeks after start of intervention.
Self-Reported Stress | At time of randomisation(March 1, 2010) and after 11 weeks
  Self-reported stress level measured using the Perceived Stress Scale-4. Questionnaire completed by participant at start and 11 weeks after start of intervention.
Self-Reported Sleep Quality | At time of randomisation(March 1, 2010) and after 11 weeks
  Self-reported sleep quality measured using the Karolinska Sleepiness Scale. Questionnaire completed by participant at start and 11 weeks after start of intervention.
Self-Reported Emotional Quality of Life | At time of randomisation(March 1, 2010) and after 11 weeks
  Self-reported emotional quality of life using the 21-Item Depression Anxiety Stress Scale, DASS-21. Questionnaire completed by participant at start and 11 weeks after start of intervention.
Self-Reported Physical Quality of Life | At time of randomisation(March 1, 2010) and after 11 weeks
  Self-reported physical quality of life measures related to urinary, bowel, and sexual function using the FACT-P questionnaire. Questionnaire completed by participant at start and 11 weeks after start of intervention.
Blodpressur, systolic and diastolic. | At time of randomisation(March 1, 2010) and after 11 weeks
  Blodpressur systolic and diastolic, will be assesed by the clinican at randomisation and after 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ove Andren, PhD, Principal Investigator — OREBRO UNIVERSITY
Locations (1):
- Orebro University, Örebro, Narke, Sweden

REFERENCES:
- [Background] Kenfield SA, Stampfer MJ, Giovannucci E, Chan JM. Physical activity and survival after prostate cancer diagnosis in the health professionals follow-up study. J Clin Oncol. 2011 Feb 20;29(6):726-32. doi: 10.1200/JCO.2010.31.5226. Epub 2011 Jan 4. PMID 21205749
- [Background] Flanagan J, Gray PK, Hahn N, Hayes J, Myers LJ, Carney-Doebbeling C, Sweeney CJ. Presence of the metabolic syndrome is associated with shorter time to castration-resistant prostate cancer. Ann Oncol. 2011 Apr;22(4):801-807. doi: 10.1093/annonc/mdq443. Epub 2010 Sep 29. PMID 20880998
- [Background] Edwards LA, Woo J, Huxham LA, Verreault M, Dragowska WH, Chiu G, Rajput A, Kyle AH, Kalra J, Yapp D, Yan H, Minchinton AI, Huntsman D, Daynard T, Waterhouse DN, Thiessen B, Dedhar S, Bally MB. Suppression of VEGF secretion and changes in glioblastoma multiforme microenvironment by inhibition of integrin-linked kinase (ILK). Mol Cancer Ther. 2008 Jan;7(1):59-70. doi: 10.1158/1535-7163.MCT-07-0329. PMID 18202010
- [Background] Giovannucci E, Rimm EB, Liu Y, Leitzmann M, Wu K, Stampfer MJ, Willett WC. Body mass index and risk of prostate cancer in U.S. health professionals. J Natl Cancer Inst. 2003 Aug 20;95(16):1240-4. doi: 10.1093/jnci/djg009. PMID 12928350
- [Background] Platz EA, Leitzmann MF, Visvanathan K, Rimm EB, Stampfer MJ, Willett WC, Giovannucci E. Statin drugs and risk of advanced prostate cancer. J Natl Cancer Inst. 2006 Dec 20;98(24):1819-25. doi: 10.1093/jnci/djj499. PMID 17179483
- [Background] Li H, Stampfer MJ, Mucci L, Rifai N, Qiu W, Kurth T, Ma J. A 25-year prospective study of plasma adiponectin and leptin concentrations and prostate cancer risk and survival. Clin Chem. 2010 Jan;56(1):34-43. doi: 10.1373/clinchem.2009.133272. Epub 2009 Nov 12. PMID 19910504
- [Background] Irwin ML, Duggan C, Wang CY, Smith AW, McTiernan A, Baumgartner RN, Baumgartner KB, Bernstein L, Ballard-Barbash R. Fasting C-peptide levels and death resulting from all causes and breast cancer: the health, eating, activity, and lifestyle study. J Clin Oncol. 2011 Jan 1;29(1):47-53. doi: 10.1200/JCO.2010.28.4752. Epub 2010 Nov 29. PMID 21115859
- [Background] Keogh JW, MacLeod RD. Body composition, physical fitness, functional performance, quality of life, and fatigue benefits of exercise for prostate cancer patients: a systematic review. J Pain Symptom Manage. 2012 Jan;43(1):96-110. doi: 10.1016/j.jpainsymman.2011.03.006. Epub 2011 Jun 2. PMID 21640547
- [Background] Tudor-Locke C, Craig CL, Brown WJ, Clemes SA, De Cocker K, Giles-Corti B, Hatano Y, Inoue S, Matsudo SM, Mutrie N, Oppert JM, Rowe DA, Schmidt MD, Schofield GM, Spence JC, Teixeira PJ, Tully MA, Blair SN. How many steps/day are enough? For adults. Int J Behav Nutr Phys Act. 2011 Jul 28;8:79. doi: 10.1186/1479-5868-8-79. PMID 21798015
- See also: Orebro University English Homepage — http://www.oru.se/English/
- See also: Harvard School of Public Health Homepage — http://www.hsph.harvard.edu/